CLINICAL TRIAL: NCT01800643
Title: Evaluation of Plasmatic Levels of Busulfan in Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Iracema Esteves, MD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Busulfan-2013
Record Dates: First submitted 2013-02-25; First posted 2013-02-28 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Acute Leukemia; Chronic Leukemia; Lymphoproliferative Disease; Myeloproliferative Disease; Immunodeficiency
Keywords: Busulfan; plasmatic dosage; Stem Cell Transplantation
MeSH Terms: conditions — Lymphoproliferative Disorders; Myeloproliferative Disorders; Immunologic Deficiency Syndromes | interventions — Transplantation; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orally Busulfan PK (Other): Evaluate the Pharmacokinetics of orally busulfan
  Interventions: Other: Analyze the pharmacokinetics of busulfan for transplantation
- Intravenously Busulfan PK (Other): Evaluate the Pharmacokinetics of intravenously busulfan
  Interventions: Other: Analyze the pharmacokinetics of busulfan for transplantation

INTERVENTIONS:
Other: Analyze the pharmacokinetics of busulfan for transplantation — Evaluate the Bu pharmacokinetics (PK) when the drug will be received by P.O or I.V and we will establish the target "Area Under Curve- AUC" based on a single daily dose (test dose) before HSCT. The test dose of orally Bu is 1 mg/Kg and the blood samples are collected and processed in time: 0h, 30 min, 1h, 1,5h, 2h, 3h, 4h, 5h and 6h after drug intake. After extraction of the plasma samples busulfan, quantitative analyzes of busulfan on human plasma will be performed by the liquid chromatograph. For the patients that will receive intravenously busulfan, the test dose is 32 mg/m2 and blood samples are collected in time: 0h, 30', 45', 1h, 2h, 3h, 4h, 5h, 6h and 8h after drug intake. The dose during the conditioning will depend on the test dose and the AUC target.
  Other Names: Busulfan dosing; Busulfan Pharmacokinetics; Busilvex; Myleran

SUMMARY:
The purpose of this prospective study is evaluate the best dose of busulfan for each patient undergoing Haematopoietic Stem Cell Transplantation

DETAILED DESCRIPTION:
* Busulfan is an alkylating antineoplastic agent used commonly during the conditioning regimen in patients undergoing Haematopoietic Stem Cell Transplantation (HSCT). Due to the fact that this drug has a variable metabolism in different individuals, the investigators performed the plasmatic dosage of chemotherapy before starting the conditioning regimen (test dose) as a way to predict the best dose to them during the conditioning. Busulfan toxicities depends on the "Area Under Curve" and Concentration Steady State (CSS).
* The investigators randomized in groups according to the route of drug administration: per oral and intravenously. Dose test will be performed before conditioning and othe pharmacokinetics (Pk) study will be made in the first day of conditioning. The test dose of P.O busulfan will be 1 mg/Kg/dose and 32 mg/m2 for I.V busulfan. The target dose of busulfan during the conditioning will depends on the Pk obtained during the test dose. In the first day of regimen, other samples will be analysed and the new AUC will be adjusted. We will have a control group who have never performed monitoring before (retrospective group)
* Test Dose for oral busulfan will be performed with peripheral blood samples at the time: 0h (before taking busulfan), 30', 1h, 1,5h, 2h, 3h, 4h, 5h and 6h. In the first day of conditioning other samples will be collected again in the same moments.
* Test dose for I.V busulfan will be performed on time 0h, 30', 45', 1h, 2h, 3h, 4h, 5h, 6h and 8h after receiving I.V busulfan. If the patients will receive I.V busulfan during conditioning, the blood samples should be collected on time 0h, 30', 1h, 2h, 3h, 4h, 5h, 6h, 7h and 8h after taking busulfan. The blood samples will be centrifuged (4º C/ 3200 rpm/10 minutes) and analysed.
* Patients will be monitored with pharmacokinetic's drug and clinical outcomes. The investigators will evaluate acute and chronic toxicities after Stem Cell Transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hematologic or non-hematologic pathology using as part of the conditioning regimen busulfan;
* Men, women and children regardless of age;
* Performance Status> 80 or ECOG <2;
* Total bilirubin <2 mg / dl and transaminases <3 times the upper limit of normal;
* Creatinine <1.5 mg / dl;
* LVEF> 50% by echocardiogram or MUGA at rest;
* Pulmonary function test with FEV1> 70%;
* Consent form signed before the start of any specific procedure.

Exclusion Criteria:

* Presence of infectious process in uncontrolled activity;
* Presence of psychiatric disorder;
* Pregnancy;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Dosing of plasmatic levels of busulfan | 2 years
  To study the effectiveness dosing of busulfan plasma levels during the administration of orally busulfan or intravenous prior to HSCT (test dose) and correlate with the respective plasma measurements in the first days of conditioning

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Evaluation of 5-years overall survival in patients who underwent different formulations of busulfan during stem Cell Transplantation
Cumulative incidence of relapse and non relapse mortality | 5 years
  Evaluate 5-years cumulative incidence of relapse and non relapse mortality in patients that underwent stem cell transplantation with busulfan in conditioning regimen
Disease Free Survival | 1 year
  Evaluate 1-year Disease Free Survival in patients that underwent stem cell transplantation with busulfan in conditioning regimen who enter complete remission after
Toxicity | 1 year
  Evaluate hematological and non hematological toxicity in patients that underwent stem cell transplantation with busulfan in conditioning regimen

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Hamerschlak, Doctor, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Esteves I, Santos FPS, Fernandes JF, Seber A, Oliveira JSR, Hamerschlak N, Kerbauy FR, S Andersson B, de Lima M. Pharmacokinetics analysis results are similar for oral compared to intravenous busulfan in patients undergoing hematopoietic stem cell transplantation, except for the earlier onset of mucositis. A controlled clinical study. Bone Marrow Transplant. 2019 Nov;54(11):1799-1804. doi: 10.1038/s41409-019-0521-5. Epub 2019 May 14. PMID 31089278